CLINICAL TRIAL: NCT06564389
Title: A PHASE 1, FIRST IN HUMAN, RANDOMIZED, DOUBLE-BLIND, SPONSOROPEN, PLACEBO-CONTROLLED, SINGLE- AND MULTIPLE DOSE ESCALATION, PARALLEL GROUP STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF PF-07832837 IN HEALTHY PARTICIPANTS AND PARTICIPANTS WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: FIH Study to Evaluate the Tolerability of PF-07832837 in Healthy Adults and Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C4991001; NCT06564389 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Atopic Dermatitis
Keywords: healthy; atopic dermatitis; first in human; monoclonal antibody; anti-inflammatory; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PF-07832837 (Experimental): single or multiple doses of PF-07832837 at ascending dose levels
  Interventions: Drug: PF-07832837
- placebo (Placebo Comparator): single or multiple doses of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-07832837 — escalated doses of PF-07832837
  Arms: PF-07832837
Other: Placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics of escalating single and repeat doses of PF-07832837 in healthy participants and in participants with moderate to severe atopic dermatitis. An additional goal is to assess the pharmacodynamics of PF-07832837 in participants with moderate to severe AD, including potential effects on clinical signs and symptoms

DETAILED DESCRIPTION:
This is a first-in-human (FIH) study of PF-07832837 that will be conducted in 2 parts: Part 1 will be conducted in healthy adult participants and Part 2 will be conducted in adult participants with moderate to severe AD.

Part 1 is within-cohort randomized, participant- and investigator-blind, sponsor-open, placebo-controlled investigation of the safety, tolerability, PK, and immunogenicity following single and multiple ascending doses of PF-07832837 in healthy participants. Part 1 may also include a cohort of Japanese healthy adult participants to provide safety, tolerability, and PK data in Japanese population to enable the inclusion of Japanese participants in future clinical trials.

Part 2 is a randomized, participant- and investigator-blind, sponsor-open, placebo-controlled study to investigate the safety, tolerability, PK, and pharmacodynamics (including clinical effects) of PF-07832837 in participants with moderate to severe AD. Part 2 will consist of cohorts of participants with moderate to severe AD. A total of approximately 28 participants will receive either active PF-07832837 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 only: Adult participants between 18 to 55 years of age, inclusive, at the time of signing the ICD
* Part 2 only: Adult participants, who at the time of screening, are between the ages of 18 and 70 years, inclusive.
* Part 1 only: Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital sign assessments, temperature, 12-lead ECGs, laboratory tests
* BMI of 17.5 to 40 kg/m2; and a total body weight >50 kg (110 lbs)
* Part 2 only: Must meet the following AD criteria:

  1. Have a clinical diagnosis of chronic AD (also known as atopic eczema) for at least 1 year prior to Day 1 and have the diagnosis of AD confirmed by photographs (at screening) and diagnostic criteria for AD.
  2. Either an inadequate response to treatment with standard of care treatments (excluding systemic immunosuppressant treatments) consistent with AD treatment guidelines (for at least 4 consecutive weeks within 6 to 12 months (depending on time since initial diagnosis) of the first dose of the study intervention. OR Have a documented reason why topical treatments are considered medically inappropriate within the last year.
  3. Have moderate to severe AD (defined as having an affected BSA (captured as part of EASI) ≥10%, IGA ≥3, and EASI ≥12 at both the screening and baseline visits).
  4. Have an otherwise healthy medical evaluation (other than signs and symptoms of AD) including medical history, physical examination, vital sign assessments, temperature, 12-lead ECGs, laboratory tests.

Controlled comorbid diseases are acceptable so long as they do not require administration of prohibited medications. This includes participants with mild or moderate asthma that is well-controlled (not requiring high dose inhaled corticosteroids, systemic [oral or parenteral] corticosteroids, or biologic asthma treatments).

Exclusion Criteria:

* Have a history of systemic infection requiring hospitalization and parenteral antimicrobial therapy, any lymphoproliferative disorder, malignancies.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, immunological/rheumatological disorder.
* Have undergone significant trauma or major surgery within 1 month of the first dose of study intervention.
* Evidence of active, latent, or inadequately treated infection with Mycobacterium tuberculosis (TB) as defined by both of the following:

  1. A positive QuantiFERON-TB Gold In-tube or equivalent test.
  2. History of either untreated or inadequately treated latent or active TB infection, or current treatment for the same.

Part 2 Only

* Currently have active forms of other inflammatory skin diseases
* Have history of or current evidence of skin conditions at the time of Day 1 that would interfere with evaluation of atopic dermatitis or response to treatment. Have active chronic or acute skin infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks prior to Day 1, or superficial skin infections within 1 week prior to Day 1.
* Score of ≥ 5 on the Fitzpatrick Skin Type Assessment.
* History of anaphylaxis with the following exceptions: participants with sensitivity and/or anaphylaxis only to a single, avoidable allergen (eg, aspirin, penicillin, sulfa drugs, nonsteroidal anti-inflammatory drugs [NSAIDs], peanuts) may be enrolled, if in the opinion of the investigator, the participant is aware of the hypersensitivity and avoids the problematic allergen. Participants must carry appropriate treatment for anaphylaxis and must know how to manage anaphylactic reactions.
* Any investigational or experimental therapy taken or procedure performed for AD, psoriasis, psoriatic arthritis, rheumatoid arthritis or other inflammatory diseases in the previous 1 year should be discussed with the Pfizer Medical Monitor (or designee).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) and serious adverse events (SAEs) Following single ascending doses (SAD) | Baseline up to Day 35
  An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or other important medical events. An AE was considered as treatment emergent if the event started during the effective duration of treatment. All events that started on or after the first dosing day up to the last dose plus the lag time were considered as TEAEs.
Number of Participants with Clinically significant Laboratory Abnormalities Following SAD | Baseline up to Day 35
  Number of participants with any laboratory test abnormalities meeting pre-defined criteria was reported in this outcome measure.
Number of Participants with Change from Baseline in Electrocardiogram (ECG) Findings Following SAD | Baseline up to Day 35
  Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR interval, QT interval, corrected QT (QTc) intervals and QRS complex. Clinically significant findings were determined by the investigator.
Number of Participants with Clinically Significant Change from Baseline in Vital Signs Following SAD | Baseline up to Day 35
  Vital signs included blood pressure, pulse rate, respiratory rate, oxygen saturation and oral temperature. Clinically significant findings were determined by the investigator.
Number of Participants with Clinically Significant Change from Baseline in Cardiac Telemetry Findings Following SAD | Day 1
  Cardiac telemetry was collected in Part 1 SAD cohorts only. Number of participants with any cardiac telemetry abnormalities were reported in this outcome measure.
Number of Participants With Treatment Emergent Treatment-Related AEs and SAEs Following multiple ascending doses (MAD) | Baseline up to Day 50
  An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or other important medical events. An AE was considered as treatment emergent if the event started during the effective duration of treatment. All events that started on or after the first dosing day up to the last dose plus the lag time were considered as TEAEs.
Number of Participants with Clinically significant Laboratory Abnormalities Following MAD | Baseline up to Day 50
  Number of participants with any laboratory test abnormalities meeting pre-defined criteria was reported in this outcome measure.
Number of Participants with Change from Baseline in Electrocardiogram (ECG) Findings Following MAD | Baseline up to Day 50
  Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR interval, QT interval, corrected QT (QTc) intervals and QRS complex. Clinically significant findings were determined by the investigator.
Number of Participants With Treatment Emergent Treatment-Related AEs and SAEs in participants with atopic dermatitis (AD) | Baseline up to Day 80
  An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose: resulted in death; required inpatient hospitalization or prolongation of existing hospitalization; was life-threatening; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or other important medical events. An AE was considered as treatment emergent if the event started during the effective duration of treatment. All events that started on or after the first dosing day up to the last dose plus the lag time were considered as TEAEs.
Number of Participants with Clinically significant Laboratory Abnormalities in participants with AD | Baseline up to Day 80
  Number of participants with any laboratory test abnormalities meeting pre-defined criteria was reported in this outcome measure.
Number of Participants with Clinically Significant Change from Baseline in Vital Signs in participants with AD | Baseline up to Day 78
  Vital signs included blood pressure, pulse rate, respiratory rate, oxygen saturation and oral temperature. Clinically significant findings were determined by the investigator.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last (AUClast) of PF-07832837 following SAD | Day 1 to Day 35
  estimated by Linear/Log trapezoidal method
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-07832837 following SAD | Day 1 to Day 35
  AUClast + (Clast*/kel), where Clast* is the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis
Maximum Observed Serum Concentration (Cmax) of PF-07832837 following SAD | Day 1 to Day 35
  Observed directly from data
Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-07832837 following SAD | Day 1 to Day 35
  Observed directly from data as time of first occurrence
Terminal serum elimination half life (t1/2) of PF-07832837 following SAD | Day 1 to Day 35
  Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the loglinear concentration time curve. Only those data points judged to describe the terminal log-linear decline will be used in the regression
Area Under the Serum Concentration-Time Curve Over the Dosing Interval (AUCtau) of PF-07832837 following MAD | Day 1 to Day 22
  Linear/log trapezoidal method
Maximum Observed Serum Concentration (Cmax) of PF-07832837 following MAD | Day 1 to Day 22
  Observed directly from data
Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-07832837 following MAD | Day 1 to Day 22
  Observed directly from data as the time of first occurrence
Percent change from baseline in Eczema Area and Severity Index (EASI) total score at Week 8 | Baseline, Week 8
  EASI evaluates severity of participants' AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4991001